CLINICAL TRIAL: NCT01564524
Title: Structural Fat Grafting for Craniofacial Trauma: Effect of Concentrating Endogenous Stromal Cells in the Fat Graft
Brief Title: Effect of Concentrating Endogenous Stromal Cells in the Fat Graft
Status: Terminated | Type: Observational
Why Stopped: Funding ended
Sponsor: University of Pittsburgh (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Other Study IDs: PRO10100293
Record Dates: First submitted 2012-03-21; First posted 2012-03-27 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Facial Injuries; Adipose Tissue
Keywords: Craniomaxillofacial (CMF) Battle-injured (BI); Facial Trauma; Fat Grafts; Autogenous Fat Transfers (AFT); Wounded warriors
MeSH Terms: conditions — Facial Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Fat graft surgical procedure — The fat graft surgical procedure will concentrate the adipose stromal cells (ASCs) in the fat graft material. A blunt tip hollow cannula is used to aspirate approximately 200-400cc of fat tissue. The aspirated fat is divided into two portions: one portion will be processed as standard graft material, the other portion will be used in a processing step that concentrates the ASCs. The aspirated fat processed as standard graft material will be divided into small alioquots and centrifuged to separate the aqueous and oil layers, and transferred into 1ml syringes. Standard fat graft material will serve as a control treatment and will be injected into one area of the face. The ASC concentrated graft material will be processed so it first separates the ASCs in a brief collagenase digestion and then resuspends the ASCs in the native fat tissue from which the stromal cells were derived. The ASC concentrated fat will be injected into another region of the face.

SUMMARY:
Traumatic facial injuries, especially those sustained in military combat, are characterized by destruction of bone and soft tissue. While the bony structures of the face can be reconstructed, it is difficult to return the soft tissue back to its original form. Many times, fat grafting, a common cosmetic and reconstructive procedure, is used in hopes of improving the soft tissue deformity. Fat grafting is a procedure in which a person's own fat is taken from areas throughout the body, usually the thighs or abdomen, with a small liposuction tube. The fat is then transferred into the area that has lost volume or fullness. The fullness of the soft tissue area may decrease over time because the transferred fat can be reabsorbed by the body. Altering the current fat grafting procedure, slightly, could lead to less reabsorption and a lasting fullness of the soft tissue area outcome of the fat graft procedure.

We are conducting this research study to help us improve the surgical treatment of people who have suffered facial soft tissue loss as a result of trauma. The goal of this research study is to see how each person's fat grafts will maintain the fat over time and to measure the quality of life during a 9 month post-surgical follow-up period. The total duration of participation is approximately 11 months.

In this study, we will concentrate the fat in the fat grafting procedure to determine whether this process will maintain the fat over time. The areas treated with enhanced fat grafts will be compared with areas treated with standard of care fat grafts. At least two areas of your face will be treated with fat grafts, (standard of care fat grafts and concentrated fat grafts).

DETAILED DESCRIPTION:
Craniofacial injuries have serious psychosocial sequele and affect quality of life. Many individuals who suffer significant facial disfigurement from injury experience psychological distress and impairment in functioning not limited to the acute phase of injury, but over a longer term period of treatment, recovery, and adjustment. Until recently, treatment of disfiguring craniofacial injuries has been mostly limited to surgical flap procedures, microsurgical tissue transfer, and implantable prostheses. However, these methods can leave conspicuous scars on the face and the donor site, and in the case of implants can lead to complications associated with foreign materials. Autologous fat grafting with minimally invasive cannulas is a procedure that has been used for decades in common plastic surgery practice for facial aesthetic procedures. This technique is also a promising treatment for soft tissue reconstruction after craniofacial trauma because the graft harvest and injection are minimally invasive. The treatment is performed by using a small liposuction cannula to aspirate fat tissue from the donor site, and then re-injecting the fat into the recipient site with specialized injection cannulas. After harvest, and prior to injection, the fat graft is subjected to a mechanical processing step to separate the aqueous layer and concentrate the adipocytes. This often takes the form of centrifugation or filtering.

The main problem with autologous fat grafting is a variable resorption of the graft volume over time. As much as 30-60% of the graft volume can diminish over time. Many variables may influence the behavior of clinical fat grafts, including harvest site, harvest technique, graft preparation, and injection technique. In our current IRB approved study on fat grafting (IRB # PRO09060101), we are seeking to accurately quantify the fat graft resorption over time following a highly standardized surgical technique. Evaluation methods include a 3D surface imaging, high resolution CT scanning, and quality of life measures. This study has enrolled and treated patients without adverse event, and the evaluation methods have been performed successfully.

In this proposed study, we plan to use essentially the same surgical procedure and evaluation methods, but with modified preparation of the fat graft. This modified preparation involves concentrating the endogenous stromal cells in the graft material in an effort to increase graft retention over time. The aspirated fat material used for fat grafting consists of mature adipocytes, a small amount of fibrous tissue, and immature adipose stromal cells. These adipose stromal cells (ASCs) are a mixed population of non-lipid laden cells that serve to turn over mature adipocytes and vascular elements. "Preadipocytes," as well as endothelial precursor cells and multilineage progenitor cells, are found. Of note, ASCs have been shown to stimulate angiogenesis when stressed under hypoxic conditions and these cells may be instrumental in healing and volume retention of fat grafts. Yoshimura, et. al. (1) found that fat aspirated with a liposuction cannula (i.e. the method of fat harvest for fat grafting) is deficient in ASCs compared to whole fat. This is due to the fact that a major portion of ASCs are located around larger blood vessels that are left intact in the donor site after liposuction with a blunt cannula.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and able to provide informed consent
2. Have suffered injury resulting in craniofacial volume defects which could be treated with a graft volume of between 3 and 100 cc of lipoaspirate
3. Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
4. Volume defects are covered by intact skin and do not communicate with oral cavity or sinuses
5. The three dimensional geometry of the volume defects would allow for treatment with lipoaspirate injection so that at least two distinct treated areas could be discerned on gross examination and radiographically (e.g. treated regions are on opposite sides of the face, on lower face versus upper face, or separated by a bony landmark such as zygoma. This would include the ability to treat an uninjured regions with fat grafts in order to obtain symmetry or balance.
6. Willing and able to comply with follow up examinations, including radiographic studies

Exclusion Criteria:

1. Age less than 18 years
2. Inability to provide informed consent
3. Craniofacial defects intended for treatment have open wounds or communicate with oral cavity or sinus (note: presence of such a defect in the setting of another defect(s) that meets treatment criteria will not exclude the patient from participating).
4. Active infection anywhere in the body
5. Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
6. Known coagulopathy
7. Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient.
8. Pregnancy
9. Diagnosis of Schizophrenia or Bipolar Disorder

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Civilian or military
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Fat grafting for facial trauma, facilitated by enhancing graft quality with a higher concentration of endogenous autologous adipose stromal cells in the grafted tissue, will enable successful restoration of tissue volume and craniofacial form. | Will take at months 9 after the fat grafting procedure
  Facial appearance and persistence of graft volume will be assessed using aesthetic grading scales, state of the art 3D photography, and high resolution CT scanning with 3D reconstruction. Subjects will be followed for 9 months after graft procedure to define long term outcomes.

SECONDARY OUTCOMES:
Measure quality of life in subjects after grafting using validated psychosocial measures. | 9 months
  A comprehensive battery of tests for evaluation of quality of life has been assembled for this study. It is important to properly determine the impact of the surgical changes and the investigators have selected Psychosocial assessment instruments to evaluate four domains: a) Satisfaction with appearance/surgical outcomes; b) Satisfaction with Medical/Health Services; c) Social Functioning, Distress, Avoidance; d) Quality of Life and General Functioning Outcomes.
Cell assessment will include adipose ASC yield, cell proliferation and characterization, capacity for adipogenic differentiation, interactions with biomaterial scaffolds that may be used in future therapies, and analysis by flow cytometry. | At the end of the 4 week observation period after entry into the study, at which time the intervention will occur and the cells will be analyzed.
  Cell assessment will include adipose ASC yield, cell proliferation and characterization, capacity for adipogenic differentiation, interactions with biomaterial scaffolds that may be used in future therapies, and analysis by flow cytometry.

CONTACTS AND LOCATIONS:
Overall Officials: J. Peter Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Yoshimura K, Sato K, Aoi N, Kurita M, Hirohi T, Harii K. Cell-assisted lipotransfer for cosmetic breast augmentation: supportive use of adipose-derived stem/stromal cells. Aesthetic Plast Surg. 2008 Jan;32(1):48-55; discussion 56-7. doi: 10.1007/s00266-007-9019-4. Epub 2007 Sep 1. PMID 17763894
- [Background] Zhu M, Zhou Z, Chen Y, Schreiber R, Ransom JT, Fraser JK, Hedrick MH, Pinkernell K, Kuo HC. Supplementation of fat grafts with adipose-derived regenerative cells improves long-term graft retention. Ann Plast Surg. 2010 Feb;64(2):222-8. doi: 10.1097/SAP.0b013e31819ae05c. PMID 20098110